CLINICAL TRIAL: NCT04488861
Title: A Feasibility Study of a Translational Research Antenatal Clinic for IVF-conceived Pregnancies: The St Mary's After Reproductive Technology (START) Clinic
Brief Title: The START Clinic: a Feasibility Study
Acronym: START
Status: Active, not recruiting | Type: Observational
Sponsor: Manchester Academic Health Science Centre (Other)
Collaborators: Academy of Medical Sciences, UK (Other); Erasmus Medical Center (Other); Tommy's (Other)
Responsible Party: Principal Investigator, Lucy Higgins, NIHR Academic Clinical Lecturer in Obstetrics, Manchester Academic Health Science Centre
Other Study IDs: NHS001747 V2.0
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Complications; IVF; Fetal Growth Retardation; Preeclampsia; Placenta Diseases
MeSH Terms: conditions — Pregnancy Complications; Fetal Growth Retardation; Pre-Eclampsia; Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood (pre-delivery) Maternal urine Maternal saliva Maternal hair Placental tissue Umbilical cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IVF-conceived: Those who have conceived by IVF (for whatever indication); target 80 participants of which it is anticipated 20 would have conceived by frozen embryo transfer IVF.
  Interventions: Other: Non-interventional cohort study
- Spontaneously conceived: Those who have conceived spontaneously (within 12 months and without use of hormonal or other contraception); target 20 participants
  Interventions: Other: Non-interventional cohort study
- Ovulation induction-conceived: Those who have conceived by ovulation induction (after more than 12 months); target 20 participants.
  Interventions: Other: Non-interventional cohort study

INTERVENTIONS:
Other: Non-interventional cohort study — Non-interventional cohort study

SUMMARY:
This is a study of the feasibility of a translational research clinic for pregnancies conceived by in vitro fertilisation (IVF). A group of at least 120 pregnancies (of which, at least 80 IVF-conceived) will be followed from early pregnancy to delivery, in order to gain early insights into the growth of the baby before birth, the physical and emotional adaptation of the mother to the pregnancy and how the placenta works. The investigators will collect preliminary data on how these factors may differ between pregnancies conceived with and without IVF, and between different IVF treatment modalities such as fresh or "frozen" embryo transfer IVF. The study aims to understand the practicalities of such a clinic, to identify barriers to participation in the clinic, to assess the uptake of different research measurements and to identify key measurements/time points with the greatest potential to identify and understand the origin of fetal growth and maternal adaptation differences after IVF conception in a full scale study.

DETAILED DESCRIPTION:
The primary objective of the study is to test the feasibility of establishing the first IVF-conceived pregnancy antenatal clinic specifically to collect longitudinal data relating to the growth of the baby in the womb, how the mother's heart and blood vessels adapt to the increased workload of pregnancy, and how the mother's emotional health (particularly stress and anxiety) varies throughout pregnancy.

The feasibility of the study protocol will be assessed using stop/go (or progression) criteria, to help determine whether future, larger scale studies of the same should be commenced. The information gathered to answer the primary and secondary outcomes of the study's primary objective will be essential for understanding, and overcoming, potential barriers to recruitment to future cohort studies within the clinic. It will enable the researchers to plan future studies with sufficient sample size to answer the specified question, realistic recruitment targets and timescales to achieve this, and using investigations that are shown to be acceptable to the majority of individuals in the target population. The secondary objective of the study is to gather preliminary data relating to the effects of fresh and frozen embryo transfer IVF on fetal, maternal and placental health.

The study is based on the design of several successful pregnancy cohort studies (such as the Tommy's Project), which run through five translational research clinics in St. Mary's Hospital, Manchester University Hospitals National Health Service (NHS) Foundation Trust: VELOCITY clinic, Lupus in Pregnancy service, Manchester Placenta Clinic, Rainbow clinic and Manchester Antenatal Vascular Service. The START clinic replicates the model of care offered through these existing clinics, offering the same levels of specialised, continuity of care to individuals who have conceived by IVF. These successful recruitment and retention within these studies gives confidence in the acceptability of the study.

The study design is a cohort study. This is where individual participants can be divided into groups by specified characteristics, in this case whether or not they had conceived by IVF or not (or sub-categorised by individual factors within the IVF treatment process, such as whether the embryo was transferred fresh or after a period of cryopreservation). No active intervention (medicine or procedure) will be administered during the study. However, it is known that health outcomes of individuals participating in research may be influenced by the experience of participating in the study itself. For this reason the investigators will also recruit "control" participants (those who have conceived without IVF, either spontaneously or with medication to aid the release of eggs, known as ovulation induction). By comparing the two groups, this will enable the research to isolate the specific effects of the IVF-conception, from the effects of being highly monitored in a research study. The investigators intend to recruit a minimum of 120 individuals across a period of three years, with approximately 4 individuals who have conceived by IVF to every 1 individual who has conceived without IVF.

Appointments in the START clinic will be arranged roughly 4-6 weekly (at approximately 9, 17, 23, 28, 33, 37 and 41 weeks). At each appointment the patient will be reviewed by a doctor and midwife from a small team of clinicians who will provide continuity of care. Routine scheduled antenatal care will be performed, along with additional measurements of fetal and placental growth and cardiovascular function, questionnaires relating to environmental exposures, modifiable risks, and emotional health, and samples of maternal blood, urine, saliva and hair. More frequent appointments will be scheduled according to local hospital guidance if complications of pregnancy are suspected or confirmed, this may mean that clinical measurements and ultrasound examinations are performed more frequently than at the planned study visits. Questionnaires and biological samples will only be administered/obtained at the (study visit closest to) stated gestational intervals. Participants will be made aware of which measurements are part of standard antenatal care and which investigations are for research; research measurements will be analysed blinded to participant identity/pregnancy outcome after conclusion of the pregnancy and will not contribute to their care during or after the pregnancy. Participants can decline particular investigations entirely or on occasion without detriment to their overall care. Where necessary, according to the individual needs of the participant, antenatal care will be shared with community midwives and other antenatal services where additional appointments are required outside the stated schedule.

At birth, the placenta and fetal blood contained within it after clamping of the umbilical cord, will be collected. Placental tissue may be used immediately after birth in experiments to study how it functions, or small amounts may be processed and stored (according to local standard operating procedures) for later assessment of its structure and functional footprint. Should histopathological examination of the placenta be indicated for clinical reasons (<5% of all pregnancies), the remaining placental tissue will be made available for this purpose according to standard local protocols for combined research and histopathological placental examination; otherwise unused placental tissue will be disposed sensitively according to local National Health Service procedures. Prior to discharge from the hospital, and preferably within 3 days of birth, the baby will be measured (using a tape measure) once for head, abdominal and thigh circumference, and length. Their skinfold thickness (to measure fat depth) over the shoulder blade and under the upper arm will be measured using purpose-built callipers. The baby will be kept warm and comfortable throughout, and the examination paused or stopped should the baby show distress, need feeding or changing or any medical intervention be required.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age at enrolment of between 18 -39 years
2. (Current pregnancy) Conception by IVF, or spontaneously ("naturally") within 12 months of trying to conceive, or with medication to stimulate egg release (ovulation induction) after a delay in conceiving of more than 12 months
3. Antenatal care and delivery planned at St. Mary's Hospital, Manchester
4. Pregnant with one, live baby within the womb (known medically as a singleton, viable, intrauterine pregnancy) at the time of recruitment
5. Able to give informed consent, with or without the use of interpretation services

Exclusion Criteria:

1. Prisoners
2. Maternal age at enrolment younger than 18 or greater than or equal to 40 years.
3. Conception in current pregnancy by non-IVF, non-Intra Cytoplasmic Sperm Injection fertility treatment (e.g. intrauterine insemination, intracervical insemination, gamete or zygote intrafallopian transfer), ovulation induction without delay in conception of at least 12 months' duration, or spontaneous conception after a delay in conception of more than 12 months, or during use of (regular or emergency hormonal or intrauterine) contraception. Conception following condom failure without emergency hormonal contraception use is not an exclusion criteria.
4. Potential participant or partner not willing to consent to disclosure of fertility treatment records to the research team
5. Antenatal care and delivery planned at another hospital
6. Pre-existing maternal medical condition requiring specialist antenatal care beyond the scope of the SMART clinic, including BMI > 35, pre-existing diabetes and hypertension
7. Miscarriage or fetal death in utero at the point of recruitment
8. Presence of detected clinically significant (as defined by clinician in charge of care) fetal abnormalities
9. Refusal of consent, including consent of the participant and any partner to access to fertility treatment records (as applicable)
10. Language barrier not overcome by telephone or video interpretation services
11. Lack of capacity to consent despite detailed explanation, ample opportunity to ask questions and time to consider options
12. Transfer of care to another hospital out of area

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant individuals, meeting the inclusion and exclusion criteria, registering for antenatal care and delivery at Manchester University Hospitals NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility: Number of referrals received | 3 years
Recruitment feasibility: Proportion of referrals eligible for recruitment | 3 years
Recruitment feasibility: Proportion of eligible individuals accepting recruitment | 3 years
Recruitment feasibility: Rate of recruitment | 3 years
Recruitment feasibility: Gestation at referral/first appointment | 3 years
Recruitment feasibility: Rate of consent to contact for future studies involving mother or child | 3 years
Protocol feasibility: Proportion of recruits completing all study visits | 3 years
Protocol feasibility: Average number of study visits required by each individual | 3 years
Protocol feasibility: Proportion of individuals accepting each type/gestation of investigation | 3 years
Protocol feasibility: Reliability of each type/gestation of investigation | 3 years
Protocol feasibility: Rate of withdrawal / loss to follow up | 3 years
Protocol feasibility: Proportion of recruits where fertility records could be accessed | 3 years
Missing data: Proportion of recruits scanned before 12 weeks' gestation | 3 years
Missing data: Proportion of missing data points for each type/gestation of investigation | 3 years
Missing data: Proportion of fertility treatment variables that could be ascertained from fertility records | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal and Fetal Health Research Centre, University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After publication of the study findings and complete anonymisation of the data, individual patient data will be deposited in an online data repository such as Mendeley Data
Supporting Information: Study Protocol, ICF
Time Frame: 3 to 5 years
Access Criteria: Open access for completely anonymised data with appropriate metadata for interpretation. Applications to access pseudonymised data may be considered in writing to the principal investigator, subject to appropriate local approvals and a data management plan that conforms to the requirements of the University of Manchester.